CLINICAL TRIAL: NCT04653454
Title: CGM Use in Hospitalized Patients With Diabetes Mellitus
Brief Title: Continuous Glucose Monitoring in Hospitalized Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian G. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-008826
Record Dates: First submitted 2020-11-06; First posted 2020-12-04 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
Keywords: CGM, Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CGM Patients (Experimental): Patients with diabetes mellitus admitted to the hospital and using a CGM will be encouraged to continue to use these devices in inpatient setting. The device alarms of high or low glucose levels will be communicated to the nursing staff.
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — CGM data will be downloaded prior to discharge and it will be compared with hospital glucometer readings taken at the same time.

SUMMARY:
The purpose of this study is to determine if patient's own Continuous Glucose Monitor (CGMs) worn in the non-ICU hospital setting have adequate accuracy for blood glucose monitoring when compared to point-of-care (POC) capillary glucose measurement, and to determine if alerts given by CGMs worn in the non-ICU hospital would prevent episodes of hyperglycemia and hypoglycemia.

DETAILED DESCRIPTION:
All patients admitted to the hospital in inpatient or observation status and having a Continuous Glucose Monitor (CGMs) attached will be screened and identified by providers and nurses. An order will be placed by providers to continue patient's home CGM use in the hospital. "CGM patient agreement" describing the hospital policy for use of CGMs will be provided to the patient for signature. Patients will be encouraged to continue to wear their CGMs in the hospital unless their presence interferes with patients' medical care. CGM presence will be recorded by nursing in patient chart under LDA (lines, drains, airway) section. Patients will be approached by the research staff and will be offered enrollment in the study. A research consent will be reviewed with patients and will be provided for signature. Patients will be asked to continue to use their home CGMs in the hospital. If CGM sensor will reach the end of life, patients have the option to place a new sensor and to follow manufacturer recommendations for calibration and setting. Patients are responsible to provide their own sensors, transmitters and readers during the hospitalization period. If it is determined that the current sensor will interfere with hospital medical and surgical care (MRI testing, procedure at the site), patients will be asked to remove the CGM sensor and transmitter. Patients will have the option to replace the sensor after the procedure if they so desire.

Patients will continue to monitor their glucose level via CGM. For flash sensors, patients will be asked to scan their sensor at least every 8 and as needed. CGMs that require calibration will be calibrated by the patients using hospital glucometer readings. .

Patients alerted by their CGM about low glucose levels or fast downward or upward trending will have to notify their nursing staff. A POC blood glucose check will be done by nursing staff to confirm the alert or the trend. Treatment decisions will be made based on POC readings.

During hospitalization patients will continue to have their blood glucose checked with POC glucometers per hospital policy.

Treatment of diabetes and the associated complications, dosing of insulin, change from PO to insulin treatment and back to PO medications during hospitalization or at discharge will be done by the admitting team with help from the inpatient Endocrinology Consultation Service.

Decisions about insulin dosing or other diabetes treatments will be made based on hospital glucometer readings, and not based on CGM readings alone.

Patients will be asked to give the research team "provider access" to their cloud CGM software, or to allow the team to download their CGM data prior to discharge if their reading devices do not automatically synchronize with the cloud software.

CGM data will be compared with POC glucometer readings obtained in the hospital at approximately the same time. Different patient variables (demographics, comorbidities, labs and vitals, administered medications) will be collected from electronic health record and will be evaluated to determine if they interfere with CGM readings. The accuracy of CGM for glucose measurement in the hospital will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or 2 Diabetes Mellitus,
* Patients 18 years of age or older,
* Patients admitted under medical or surgical services.
* Patients treated with diet alone, insulin (SQ, insulin pump) or oral hypoglycemic medications.
* Have their own Continuous Glucose Monitoring (CGM) monitor present on admission or able to be placed after admission.

Exclusion Criteria:

* Individuals under 18 years of age.
* COVID-19 infection.
* Infection of the skin at the CGM site requiring removal of the sensor.
* Patients with altered Mental Status.
* Patients unable to scan their flash CGMs at least every 8 hours.
* Inability to provide written consent.
* Hospitalized for less than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20508009

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Patients: Patients with diabetes mellitus admitted to the hospital and using a CGM were encouraged to continue to use these devices in inpatient setting. The device alarms of high or low glucose levels were communicated to the nursing staff.
  Continuous Glucose Monitor (CGM): CGM data was downloaded prior to discharge and it was compared with hospital glucometer readings taken at the same time.
Period: Overall Study
Arm/Group | CGM Patients
Started | 142
Completed | 101
Not Completed | 41
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 40

BASELINE CHARACTERISTICS:
Arm/Group | CGM Patients
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.97 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 135
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 112
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitors (CGM) Accuracy - Mean Absolute Relative Difference (MARD)
Description: The absolute relative difference (ARD) was defined as the absolute difference between control - point of care (POC) glucose reading and the corresponding CGM reading divided by POC glucose reading and expressed as percentage. ARD was calculated as mean absolute relative difference (MARD) with standard deviation. MARD was calculated between matched pairs of POC (point of care) glucose readings and the closest CGM reading. MARD was summarized as mean (standard deviation) or median (range) for glucose readings <70 mg/dl, 70-180 mg/dL, >180 mg/dl, 181-250mg/dl, >250 mg/dl respectively.
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Population: 3316 total CGM-POC readings pairs were collected. Those 3316 POC-CGM reading pairs were further broken down into the following categories based on the POC value: CGM-POC Pairs with POC<70 mg/dL, CGM-POC Pairs with POC between 70-180 mg/dL, CGM-POC Pairs with POC between 181-250mg/dl, CGM-POC Pairs with POC>250 mg/dl, respectively.
Measure: Mean (Standard Deviation); unit: MARD percentage
Units Other Than Participants: CGM-POC pairs
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Number analyzed (CGM-POC pairs) | 3316
MARD percentage
  MARD for CGM-POC pairs with POC <70 mg/dL: number analyzed (CGM-POC pairs) | 106
  MARD for CGM-POC pairs with POC <70 mg/dL | 22.6 (19.5)
  MARD for CGM-POC pairs with POC between 70-180 mg/dL: number analyzed (CGM-POC pairs) | 2058
  MARD for CGM-POC pairs with POC between 70-180 mg/dL | 14.6 (12.8)
  MARD for CGM-POC pairs with POC between 181-250 mg/dL: number analyzed (CGM-POC pairs) | 757
  MARD for CGM-POC pairs with POC between 181-250 mg/dL | 11.7 (10.1)
  MARD for CGM-POC pairs with POC>250 mg/dL: number analyzed (CGM-POC pairs) | 395
  MARD for CGM-POC pairs with POC>250 mg/dL | 10.4 (8.7)
  MARD for all CGM-POC pairs | 13.7 (12.3)

2. Secondary Outcome: CGM Recorded Hypoglycemia Episodes
Description: The incidence of hypoglycemic episodes
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: Hypoglycemic Episodes
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Hypoglycemic Episodes
  Hypoglycemic Episodes <54 mg/dL | 0.47 (1.94)
  Hypoglycemic Episodes <70 mg/dL | 1.45 (3.33)
Statistical Analysis 1: Comparison: CGM Patients; Test type: Superiority; p = 0.129, Wilcoxon (Mann-Whitney) — Hypoglycemic Episodes <54 mg/dL
Statistical Analysis 2: Comparison: CGM Patients; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney) — Hypoglycemic Episodes <70 mg/dL

3. Secondary Outcome: CGM Recorded Duration of Hypoglycemic Episodes
Description: CGM recorded duration of hypoglycemic episodes
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Minutes
  Hypoglycemic Episodes <54 mg/dL | 37.810 (191.77)
  Hypoglycemic Episodes <70 mg/dL | 162.81 (572.29)
Statistical Analysis 1: Comparison: CGM Patients; Test type: Superiority; p = 0.203, Wilcoxon (Mann-Whitney) — Hypoglycemic Episodes <54 mg/dL
Statistical Analysis 2: Comparison: CGM Patients; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Hypoglycemic Episodes <70 mg/dL

4. Secondary Outcome: CGM Recorded Hyperglycemic Episodes
Description: The incidence of hyperglycemic episodes
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: Hyperglycemic Episodes
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Hyperglycemic Episodes
  Hyperglycemic Episodes >180 mg/dL | 10.216 (12.794)
  Hyperglycemic Episodes >250 mg/dL | 5.935 (8.958)

5. Secondary Outcome: CGM Recorded Duration of Hyperglycemic Episodes
Description: The duration of hyperglycemic episodes
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Minutes
  Hyperglycemic Episodes >180 mg/dL | 2419.44 (2804.85)
  Hyperglycemic Episodes >250 mg/dL | 801.99 (1171.28)
Statistical Analysis 1: Comparison: CGM Patients; Test type: Superiority; p = 0.076, Wilcoxon (Mann-Whitney) — Hyperglycemic Episodes >180 mg/dL
Statistical Analysis 2: Comparison: CGM Patients; Test type: Superiority; p = 0.038, Wilcoxon (Mann-Whitney) — Hyperglycemic Episodes >250 mg/dL

6. Secondary Outcome: Variation in Mean Absolute Relative Difference (MARD) in Relation to Pharmacological and Physiological Parameters
Description: The correlation between MARD point of care (POC) and Creatinine, Glomerular Filtration Rate (GFR), Bicarbonate, Hemoglobin (Hb), Mean Arterial Pressure (MAP), and Peripheral Oxygen Saturation (SpO2). The Spearman's rank correlation method was used to calculate the correlation coefficient.
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Number; unit: Correlation Coefficient
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Correlation Coefficient
  Creatinine | -0.08
  139GFR | -0.02
  Bicarbonate | 0.024
  Hb | -0.012
  MAP | 0.003
  SpO2 | 0.034
Statistical Analysis 1: Comparison: CGM Patients; Test type: Superiority; p < 0.0001, Spearman Correlation coefficients — Creatinine
Statistical Analysis 2: Comparison: CGM Patients; Test type: Superiority; p = 0.0002, Spearman Correlation coefficients — 139GFR
Statistical Analysis 3: Comparison: CGM Patients; Test type: Superiority; p = 0.22, Spearman Correlation coefficients — Bicarbonate
Statistical Analysis 4: Comparison: CGM Patients; Test type: Superiority; p = 0.48, Spearman Correlation coefficients — Hemoglobin
Statistical Analysis 5: Comparison: CGM Patients; Test type: Superiority; p = 0.77, Spearman Correlation coefficients — MAP
Statistical Analysis 6: Comparison: CGM Patients; Test type: Superiority; p = 0.0516, Spearman Correlation coefficients — SpO2

7. Secondary Outcome: In Hospital Mortality
Description: Mortality during index hospitalization
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Participants | 2

8. Secondary Outcome: Hospitalization Length of Stay
Description: Duration of hospital stay in hours
Time Frame: From date of enrollment and until discharge from the hospital up to 30 days.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Hours | 116.5 [74.73 to 215.43]

9. Secondary Outcome: Mortality Rate at 30 Days
Description: Mortality rate at 30 days post discharge from the hospital
Time Frame: From date of enrollment up to 60 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Participants | 0

10. Secondary Outcome: Number of Re-hospitalization Events at the Same Institution Within 30 Days From the Discharge Date of the Preceding Admission.
Description: Number of re-hospitalization events that occurred at the same institution within 30 days from the discharge date of the preceding admission.
Time Frame: From date of enrollment up to 60 days.
Measure: Count of Units; unit: Hospitalizations Events
Units Other Than Participants: Hospitalizations Events
Arm/Group | CGM Patients
Number analyzed (Participants) | 101
Number analyzed (Hospitalizations Events) | 188
Hospitalizations Events | 60

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through end of study participation, approximately 60 days.
Arm/Group | CGM Patients
All-Cause Mortality (participants affected / at risk) | 2/142
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04653454/Prot_SAP_000.pdf